CLINICAL TRIAL: NCT01115608
Title: Development of a Standardized Clinical Pharmacist Service for Patients Discharged From Hospital. Measurement of Drug Prescribing Quality in Secondary Prevention of Coronary Heart Disease Utilizing a Medication Assessment Tool (MAT-CHDsp)
Brief Title: Pharmaceutical Follow-up of Coronary Heart Disease (CHD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pharmacy of North Norway Trust (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Beate Hennie Garcia, PhD, Associate Professor, Hospital Pharmacy of North Norway Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHAN-001
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Coronary Heart Disease
Keywords: Preventive Health Services
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist follow-up (Experimental): The patients will receive pharmaceutical follow-up during one year after discharge from the hospital. Three meetings are arranged, one at discharge, one after three months and the last after one year. Patients will be called up for arrangement of "consultation". Written information concerning drugs used will be supplied.
  Interventions: Other: Pharmacist follow-up
- Control group (No Intervention): The control group receives no follow-up from the pharmacist, but will after one year, when they are out of the study, receive one follow-up visit and drug review.

INTERVENTIONS:
Other: Pharmacist follow-up — Drug review, drug conversation and written drug information. Follow-up concerning therapeutic goals and cooperation with the patient and the patient's GP to achieve these.
  Arms: Pharmacist follow-up

SUMMARY:
Objectives To explore the impact of a clinical pharmacist-led 12 month lasting follow-up program for patients with established coronary heart disease (CHD) discharged from the North Norway University Hospital. Methods A total of 102 patients aged 18-82 years were enrolled in a non-blinded, randomized controlled trial. The intervention comprised medication reconciliation, medication review and patient education during three meetings; at discharge, after three months and after twelve months. The control group received standard care from their general practitioner. Primary outcomes were adherence to clinical guideline recommendations concerning prescription, therapy goal achievement and lifestyle education defined in the medication assessment tool for secondary prevention of CHD (MAT-CHDSP). Secondary outcomes included changes in the biomedical risk factors cholesterol, blood pressure and blood glucose. Key findings Ninety-four patients completed the trial, 48 intervention group patients and 46 controls.

Appropriate prescribing was high, but therapy goal achievement was low in both study groups throughout the study. Overall adherence to MAT-CHDSP criteria increased in both groups and was significantly higher in the intervention group at study end compared to the control group, 78.1% vs. 61.4%, P < 0.001. The difference was mainly due to an increased documentation of lifestyle advices in intervention group patients.

No significant improvements in biomedical risk factors were observed in favor of the intervention group, possible due to an underpowered study. Conclusion The clinical pharmacist-led follow-up program significantly increased documented lifestyle advices defined in the MAT-CHDSP for the intervention group, but did not lead to significant improvements in biomedical risk factor measures in favor of the intervention group. Even if prescribing was high, therapy goal achievement was low in both study groups. Changes to the follow-up program are warranted, in addition to a larger, adequately powered study, before implementation in standard patient care can be recommended.

DETAILED DESCRIPTION:
Find published article in Pharm Pract (Granada). 2015 Apr-Jun; 13(2): 575. https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4482847/pdf/pharmpract-13-575.pdf

ELIGIBILITY:
Inclusion Criteria:

* established coronary heart disease
* age 18 - 80 years
* patients living in the three nearby communities Tromsoe, Balsfjord and Karlsoey, this because they need to see the pharmacist personally.

Exclusion Criteria:

* patients living in nursing homes
* patients included in NORstent, another trial including patients at the same department
* patients already receiving pharmaceutical follow-up elsewhere
* cancer patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to MAT-CHDsp (medication assessment tool based on guideline recommendations) | At baseline (both arms)
  MAT-CHDsp includes 20 review criteria assessing both appropriateness of drug prescribing, appropriateness of dose adjustments/change of drugs and appropriateness of information concerning life-style modifications. Achievment of therapeutic goals concerning lipids, blood pressure and blood glucose is also measured.
Adherence to MAT-CHDsp (medication assessment tool based on guideline recommendations) | After one year (both arms)
  MAT-CHDsp includes 20 review criteria assessing both appropriateness of drug prescribing, appropriateness of dose adjustments/change of drugs and appropriateness of information concerning life-style modifications. Achievment of therapeutic goals concerning lipids, blood pressure and blood glucose is also measured.

SECONDARY OUTCOMES:
Drug related problems | At inclusion, after three months and after one year.
  Medication reviews often reveals safety issues concerning the drug regime, except from the primary outcome measures. THese are noted and will be assessed and tried solved during follow-up in close cooperation with the GP.
Hospitalisation | After one year
  Data will be collected, both for the study group and for the control group, concerning hospitalisation during the year included in the study. The groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Trude Giverhaug, Dr.Scient., Study Chair — Hospital Pharmacy of North Norway Trust
Locations (1):
- Hospital Pharmacy of North Norway Trust, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- See also: Published Article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4482847/pdf/pharmpract-13-575.pdf